CLINICAL TRIAL: NCT05395117
Title: A Fixed Sequence, Open-label Study to Assess the Effect of Multiple Doses of AZD5462 on the Pharmacokinetics of Oral Midazolam (CYP3A4 Probe), Rosuvastatin (OATP1B1/3, BCRP Probe), and Digoxin (P-gp Probe) in Healthy Participants
Brief Title: A Study to Assess the Effect of AZD5462 on the Pharmacokinetics of Midazolam, Rosuvastatin and Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9090C00003
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Healthy Participants
Keywords: Cytochrome P450 enzyme 3A4; Organic Anion Transporting Polypeptide 1B1/1B3; Breast Cancer Resistance Protein; P-glycoprotein
MeSH Terms: interventions — Midazolam; Rosuvastatin Calcium; Digoxin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A: High dose (Experimental): Participants will receive the Investigational Medicinal Product (IMP), AZD5462 Dose A starting on Day 6 and continued until Day 18 and the following approved medicinal products:
  * Midazolam
  * Rosuvastatin
  * Digoxin
  Interventions: Drug: AZD5462; Drug: Midazolam; Drug: Rosuvastatin; Drug: Digoxin
- Treatment Arm B: Low dose (Experimental): Participants will receive the IMP, AZD5462 Dose B starting on Day 6 and continued until Day 18 and the following approved medicinal products:
  * Midazolam
  * Rosuvastatin
  * Digoxin
  Interventions: Drug: AZD5462; Drug: Midazolam; Drug: Rosuvastatin; Drug: Digoxin

INTERVENTIONS:
Drug: AZD5462 — Treatment Arm A: Participants will receive the IMP, AZD5462 Dose A starting on Day 6 and continued until Day 18 and the following approved medicinal products:
  * Midazolam
  * Rosuvastatin
  * Digoxin
  Treatment Arm B: Participants will receive the IMP, AZD5462 Dose B starting on Day 6 and continued until Day 18 and the following approved medicinal products:
  * Midazolam
  * Rosuvastatin
  * Digoxin
Drug: Midazolam — Participants will receive a single dose of midazolam in the morning of Day 1 and in the morning of Day 15 in both the arms.
Drug: Rosuvastatin — Participants will receive rosuvastatin as a single dose administered with digoxin at the same time in the morning of Day 2, Day 6, and in the morning of Day 16 in both the arms.
Drug: Digoxin — Participants will receive digoxin as a single dose administered with rosuvastatin at the same time in the morning of Day 2, Day 6, and in the morning of Day 16 in both the arms.

SUMMARY:
This study will assess the effect of multiple doses of AZD5462 on the PK of oral midazolam (CYP3A4 probe), rosuvastatin (OATP1B1/3, BCRP probe), and digoxin (P-gp probe) in healthy participants.

This study will consist of 2 treatment arms (Treatment Arms A and B) and within each treatment arm, the participants will first be administered the probe substrates (midazolam, rosuvastatin, and digoxin) alone followed by administration of the probe substrates together with AZD5462. The treatment arms differ in the dose of AZD5462 being administered and will be performed sequentially starting with Treatment Arm A (AZD5462 Dose A, high dose treatment arm) and followed by Treatment Arm B (AZD5462 Dose B, low dose treatment arm). Each treatment arm will include 5 periods.

Thirty two participants in total (16 participants per treatment arm) will be enrolled to ensure at least 24 evaluable participants (12 participants per treatment arm) at the end of the last treatment period.

A follow-up visit at Day 24 (+-1 Day) will be conducted via a phone call.

DETAILED DESCRIPTION:
This is a phase I, single-centre, 2-treatment arm, 5-period, fixed sequence study.

The Study Will Comprise of a Screening Period and Five Treatment Periods:

* Screening Period (Maximum 28 Days) Participant eligibility will be confirmed during the Screening Visit.
* Period 1 (Day 1) Single dose administration of midazolam on Day 1.
* Period 2 (Day 2) Single dose administration of rosuvastatin and digoxin on Day 2. There will be a minimum washout period of 3 days between Period 2 and Period 3.
* Period 3 (Days 6 to 14) Single dose administration of rosuvastatin and digoxin together with AZD5462 (Treatment Arm A, Dose A; Treatment Arm B, Dose B) on Day 6. AZD5462 will continue to be administered throughout the period including Day 14.
* Period 4 (Day 15) Single dose administration of midazolam together with AZD5462 (Treatment Arm A, Dose A; Treatment Arm B, Dose B) at steady state on Day 15.
* Period 5 (Days 16 to 18) Single dose administration of rosuvastatin and digoxin together with AZD5462 (Treatment Arm A, Dose A; Treatment Arm B, Dose B) at steady state on Day 16. AZD5462 will continue to be administered on Days 17 and 18.

Participants will be resident in the study centre when dosed with probe substrates (midazolam, rosuvastatin, and digoxin) and/or AZD5462 including the washout period between Period 2 and Period 3. Residency will commence on Day -1 and end on Day 20.

A follow-up visit at Day 24 (+-1 Day) will be conducted via a phone call.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and female participants aged 18 to 55 years with suitable veins for cannulation or repeated venepuncture.
* Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of non childbearing potential confirmed at screening.
* Have a Body Mass Index (BMI) between 18 and 32 kg/m2 inclusive and weigh at least 50 kg and no more than 105 kg inclusive at screening.
* Male subject must adhere to the contraception methods details.

Exclusion Criteria:

* History of any clinically significant disease or disorder which may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study including but not limited to:

  (i) Systemic sclerosis (ie, scleroderma). (ii) Moderate to severe valvular disease. (iii) Hypertrophic obstructive cardiomyopathy. (iv) Restrictive cardiomyopathy. (v) Gilbert's syndrome. (vi) History of vascular or left ventricular aneurysms or prior dissections. (vii) Any history of joint hypermobility, Marfan's Syndrome, or any connective tissue disorder.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMPs.
* Any laboratory values with deviations at screening or admission to the study centre.
* Any clinically significant abnormalities in clinical biochemistry, haematology, or urinalysis results.
* Any clinically significant abnormal findings in vital signs after 5 minutes supine rest.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12-lead ECG.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
* Known or suspected history of drug abuse.
* Has received another new chemical entity within 3 months of the first administration of IMP in this study.
* Plasma donation within 1 month of screening or any blood donation/loss > 500 mL during the 3 months prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5462.
* Current smokers or those who have smoked or used nicotine products within the 3 months prior to screening.
* Positive screen for drugs of abuse or cotinine at screening or on each admission to the study centre or positive screen for alcohol on admission to the study centre prior to the first administration of the IMP.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of any prescribed or non prescribed medication including antacids, analgesics, herbal remedies, megadose vitamins and minerals during the 2 weeks or 5 half-lives of the medication, whichever is longer, prior to the first administration of IMP.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* Excessive intake of caffeine-containing drinks or food.
* Involvement of any AstraZeneca, Parexel, or study centre employee or their close relatives.
* Participants who have previously received AZD5462.
* Participants who are vegans or have medical dietary restrictions.
* Vulnerable participants.
* Participants who cannot communicate reliably with the Principal Investigator (PI).
* Clinical signs and symptoms consistent with COVID-19 by appropriate laboratory test within the last 4 weeks prior to screening or on admission.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-versus-time curve from pre-dose (time 0) extrapolated to infinite time (AUCinf) | Midazolam: Period 1 (Day 1), and Period 4 (Day 15); Rosuvastatin and Digoxin: Period 2 (Day 2), Period 3 (Days 6 - 14), and Period 5 (Days 16 - 18)
  The effect of AZD5462 on the AUCinf of oral midazolam, rosuvastatin, and digoxin will be assessed.
Area under the concentration-versus-time curve from pre-dose (time 0) to the time of the last quantifiable concentration (AUClast) | Midazolam: Period 1 (Day 1), and Period 4 (Day 15); Rosuvastatin and Digoxin: Period 2 (Day 2), Period 3 (Days 6 - 14), and Period 5 (Days 16 - 18)
  The effect of AZD5462 on the AUClast of oral midazolam, rosuvastatin, and digoxin will be assessed.
Maximum observed serum (peak) drug concentration [Cmax] | Midazolam: Period 1 (Day 1), and Period 4 (Day 15); Rosuvastatin and Digoxin: Period 2 (Day 2), Period 3 (Days 6 - 14), and Period 5 (Days 16 - 18)
  The effect of AZD5462 on the Cmax of oral midazolam, rosuvastatin, and digoxin will be assessed.

SECONDARY OUTCOMES:
Time to reach peak or maximum observed concentration or response following drug administration (tmax) | Midazolam: Period 1 (Day 1), and Period 4 (Day 15); Rosuvastatin and Digoxin: Period 2 (Day 2), Period 3 (Days 6 - 14), and Period 5 (Days 16 - 18)
  The effect of AZD5462 on the tmax of oral midazolam, rosuvastatin, and digoxin will be assessed.
Half life associated with terminal slope (λz) of a semi logarithmic concentration time curve (t1/2λz) | Midazolam: Period 1 (Day 1), and Period 4 (Day 15); Rosuvastatin and Digoxin: Period 2 (Day 2), Period 3 (Days 6 - 14), and Period 5 (Days 16 - 18)
  The effect of AZD5462 on the t1/2λz of oral midazolam, rosuvastatin, and digoxin will be assessed.
Partial area under the serum concentration time curve from time 0 to time 12 (AUC0-12h) | Day 6, and Day 16
  The AUC0-12h of AZD5462 will be determined.
Maximum observed serum (peak) drug concentration [Cmax] | Day 6, and Day 16
  The Cmax of AZD5462 will be determined.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) | Day 6, and Day 16
  The tmax of AZD5462 will be determined.
Trough plasma exposure of AZD5462 (Ctrough) | Days 14 to 15, and Days 17 to 18
  Ctrough values of AZD5462 will be determined.
Incidence of Adverse Events (AEs) | From screening (Day -28 to Day -2) to follow-up (Day 20)
  The safety and tolerability of AZD5462 alone and in combination with midazolam, rosuvastatin, and digoxin will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home